CLINICAL TRIAL: NCT05984160
Title: Efficacy and Safety of Paragastric Neural Block in Controlling Pain, Nausea and Vomiting After Laparoscopic Sleeve Gastrectomy; Prospective Randomized Controlled Double-blind Study
Brief Title: Efficacy of Paragastric Neural Block Procedure on Postoperative Pain in Patients Who Underwent Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-22686390-050.99-27043
Record Dates: First submitted 2023-07-18; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Post Operative Pain
Keywords: Obesity; Post operative pain; Pain block; Sleeve gastrectomy
MeSH Terms: conditions — Obesity; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups as perigastric neural block and control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization was performed by a general surgeon who would not be present during the block procedure. Patients were numbered sequentially according to the randomization scheme. Patient numbers were recorded in the follow-up files. Evaluation of the postoperative results was done by a general surgeon who was unaware of the group distributions. Since both the patients and the general surgeon who will make the evaluation did not know whether the block procedure was applied or not, the study was performed as double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paragastric neural block (Active Comparator): Patients who were operated for sleeve gastrectomy were included in the study. Afterwards, they were divided into two groups. While pragastric neural block was applied to one group, no intervention was made to the other group.
  Interventions: Other: Paragastric neural block
- Control (No Intervention): Control grup

INTERVENTIONS:
Other: Paragastric neural block — A block method used to control patients' symptoms of pain, nausea and vomiting after surgery.
  Arms: Paragastric neural block

SUMMARY:
Surgical treatment is the most effective way to achieve effective and sustainable weight loss in patients with obesity and to improve the comorbidities caused by it.

Although minimally invasive bariatric surgical procedures are applied today, postoperative pain is one of the most basic problems. Opioid-derived drugs used for pain control cause respiratory depression and constipation. Enhanced Recovery After Surgery (ERAS) protocols recommend reducing opioid use after bariatric surgery to help patients have a healthier postoperative period.

Different methods such as transversus abdominis plane (TAP) block and erector spinae plane (ESP) block are used to reduce the postoperative opioid dose and for effective pain control. While these methods are effective in controlling somatic pain, they have no effect on visceral pain.

It has been shown that patients' pain and opioid consumption decrease especially after celiac plexus block. Vagal and sympathetic afferent stimuli from the gastrointestinal tract, on the other hand, stimulate the vomiting center and cause nausea and vomiting. Paragastric neural block is a new method performed by injecting local anesthetic into the posterosuperior paragastric area in the area covering the left gastric artery by revealing the esophagogastric junction, proximal stomach, middle of the stomach, distal antrum, hepatoduodenal ligament and stomach posterior along the border of the lesser omentum. In this way, it is aimed to prevent both visceral pain and the symptoms of nausea and vomiting.

In our study, the investigators aimed to evaluate the efficacy and safety of paragastric nerve block applied during laparoscopic sleeve gastrectomy by comparing it with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of over 35 and an obesity-related comorbidity,
* Body mass index of over 40,
* Patients who underwent laparoscopic sleeve gastrectomy,
* ASA risk score of 2-3,
* Agreed to be included in the study.

Exclusion Criteria:

* Chronic pain disorder or using gabapentin,
* Opioid addicts,
* Using anticoagulant drugs,
* History of previous upper gastrointestinal system surgery,
* Surgical complications during or after surgery,
* Hepatic or renal failure,
* Moderate or severe cardiovascular or respiratory disease,
* Allergy to the local anesthetic agent to be applied for the block,
* Limited cooperation,
* More than one surgical intervention in the same session,
* Allergy to the drugs to be used in the postoperative treatment protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | In first 24 hours
  The investigators used visual analog scale. Minimum value 0 (means no pain), maximum values 10 (means worst pain ever).
Postoperative nause and vomiting | In first 24 hours
  The investigators used Post operative nause and vomiting impact scale. Minimum value 0, maximum values 6. Total score >4 defines clinically important postoperative nause and vomiting.

SECONDARY OUTCOMES:
First Rescue analgesia | In first 24 hours
  Did patients need first rescue analgesia?
Second Rescue analgesia | In first 24 hours
  Did patients need second rescue analgesia?
Rescue antiemetic | In first 24 hours
  Did patients need rescue antiemetic drug?
Time to rescue antiemetic | In first 24 hours
  When patients need rescue antiemetic drug?
Time to first rescue analgesia | In first 24 hours
  When patients need first rescue analgesia?
Time to second rescue analgesia | In first 24 hours
  when patients need second rescue analgesia?
First mobilization time | In first 24 hours
  When patients start to walk?
Operation time | Through operation completion, an avarage of 1 hour
  How long did the surgery take?
Patient satisfaction | In first 72 hours
  The investigators used likert scale. Minimum value 1 (very unsatisfied), maximum values 5 (very satisfied).
Pulse before block | at block moment
  Pulse before block
Pulse 10 minutes after the block | 10 minutes after the block
  Pulse 10 minutes after the block
Sistolic blood pressure before the block | at block moment
  Sistolic blood pressure before the block
Sistolic blood pressure 10 minutes after the block | 10 minutes after the block
  Sistolic blood pressure 10 minutes after the block
Diastolic blood pressure before the block | at block moment
  Diastolic blood pressure before the block
Diastolic blood pressure 10 minutes after the block | 10 minutes after the block
  Diastolic blood pressure 10 minutes after the block
Complication at the block site | Through operation, an avarage of 1 hour
  Were there any complications during the block?

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet K Katar, Assoc.Prof., Principal Investigator — Atlas University
Locations (1):
- Atlas university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the article is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start after the publication.
Access Criteria: All results of working can be shared with researchers after the study is published.

REFERENCES:
- [Background] Peeters A, Barendregt JJ, Willekens F, Mackenbach JP, Al Mamun A, Bonneux L; NEDCOM, the Netherlands Epidemiology and Demography Compression of Morbidity Research Group. Obesity in adulthood and its consequences for life expectancy: a life-table analysis. Ann Intern Med. 2003 Jan 7;138(1):24-32. doi: 10.7326/0003-4819-138-1-200301070-00008. PMID 12513041
- [Background] Arterburn DE, Olsen MK, Smith VA, Livingston EH, Van Scoyoc L, Yancy WS Jr, Eid G, Weidenbacher H, Maciejewski ML. Association between bariatric surgery and long-term survival. JAMA. 2015 Jan 6;313(1):62-70. doi: 10.1001/jama.2014.16968. PMID 25562267
- [Background] Liu JJ, Brenner DM. Opioid-Related Constipation. Gastroenterol Clin North Am. 2022 Mar;51(1):107-121. doi: 10.1016/j.gtc.2021.10.007. Epub 2022 Jan 8. PMID 35135657
- [Background] Budiansky AS, Margarson MP, Eipe N. Acute pain management in morbid obesity - an evidence based clinical update. Surg Obes Relat Dis. 2017 Mar;13(3):523-532. doi: 10.1016/j.soard.2016.09.013. Epub 2016 Sep 19. PMID 27771314
- [Background] Stenberg E, Dos Reis Falcao LF, O'Kane M, Liem R, Pournaras DJ, Salminen P, Urman RD, Wadhwa A, Gustafsson UO, Thorell A. Guidelines for Perioperative Care in Bariatric Surgery: Enhanced Recovery After Surgery (ERAS) Society Recommendations: A 2021 Update. World J Surg. 2022 Apr;46(4):729-751. doi: 10.1007/s00268-021-06394-9. Epub 2022 Jan 4. PMID 34984504
- [Background] Emile SH, Abdel-Razik MA, Elbahrawy K, Elshobaky A, Shalaby M, Elbaz SA, Gado WA, Elbanna HG. Impact of Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Pain and Early Outcome After Laparoscopic Bariatric Surgery: a Randomized Double-Blinded Controlled Trial. Obes Surg. 2019 May;29(5):1534-1541. doi: 10.1007/s11695-019-03720-y. PMID 30706309
- [Background] Zengin SU, Ergun MO, Gunal O. Effect of Ultrasound-Guided Erector Spinae Plane Block on Postoperative Pain and Intraoperative Opioid Consumption in Bariatric Surgery. Obes Surg. 2021 Dec;31(12):5176-5182. doi: 10.1007/s11695-021-05681-7. Epub 2021 Aug 27. PMID 34449029
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617
- [Background] Kambadakone A, Thabet A, Gervais DA, Mueller PR, Arellano RS. CT-guided celiac plexus neurolysis: a review of anatomy, indications, technique, and tips for successful treatment. Radiographics. 2011 Oct;31(6):1599-621. doi: 10.1148/rg.316115526. PMID 21997984
- [Background] Rana MV, Candido KD, Raja O, Knezevic NN. Celiac plexus block in the management of chronic abdominal pain. Curr Pain Headache Rep. 2014 Feb;18(2):394. doi: 10.1007/s11916-013-0394-z. PMID 24414338